CLINICAL TRIAL: NCT05297175
Title: Feasibility of the Trammpolin® Medial Meniscus Prosthesis Intended to Restore the Medial Meniscus Function to Provide Pain Relief After Meniscectomy
Brief Title: AIR (Artificial Implant to Restore the Medial Meniscus Function)2 Clinical Investigation
Acronym: AIR2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: ATRO Medical B.V. (Industry)
Collaborators: Avania (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AM-002
Record Dates: First submitted 2022-02-14; First posted 2022-03-28 (Actual); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: Knee Injuries and Disorders
Keywords: Medial meniscus prosthesis; Symptomatic uni-compartmental pain
MeSH Terms: conditions — Knee Injuries; Disease

STUDY DESIGN:
Intervention Model Description: Early feasibility study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Other): Implantation of a medial meniscus prosthesis in the medial knee compartment of a post medial meniscectomy knee.
  Interventions: Device: Trammpolin medial meniscus prosthesis

INTERVENTIONS:
Device: Trammpolin medial meniscus prosthesis — Implantation of the Trammpolin medial meniscus prosthesis in patients with a severe medial meniscus damage

SUMMARY:
The AIR2 Study is a multi-center, prospective, interventional clinical trial with the objective to evaluate the safety and performance of the Trammpolin® medial meniscus prosthesis.

DETAILED DESCRIPTION:
The Trammpolin® meniscus prosthesis is intended to replace the native medial meniscus to provide pain relief in the medial compartment of the knee joint, when this is caused by medial partial meniscectomy.

Patients who meet the inclusion/exclusion criteria and who are implanted with the Trammpolin® medial meniscus prosthesis will be followed for 2 years. The patient reported outcome measures for knee pain and function, and knee clinical condition by MRI and X-ray is assessed post-operative compared to pre-operative.

ELIGIBILITY:
Inclusion Criteria:

1. Has medial compartment knee pain and had a medial partial or total meniscectomy > 6 months ago. The lack of meniscus tissue is confirmed by patient history and MRI
2. Has a KOOS Pain of ≤ 75 (100 being no pain and the highest attainable score)
3. Is between age 18 and 70 years (inclusive) at the time of screening
4. Has neutral alignment ± 5° of the mechanical axis, i.e., the angle formed by a line drawn from the center of the femoral head to the medial tibial spine and a line drawn from the medial tibial spine to the center of the ankle joint, as confirmed by X-ray
5. Is willing to be implanted with the Trammpolin® medial meniscus prosthesis
6. Is willing and able to comply to the clinical investigation required follow up visits, questionnaires, X-rays and MRI's
7. Is able and willing to understand and sign the clinical investigation Informed Consent Form
8. Is able to read and understand the national language of the country in which the relevant clinical site is located

Exclusion Criteria:

1. Has a symptomatic knee because of a tear that could potentially be addressed by a repeat partial meniscectomy
2. Has evidence of a modified Outerbridge Grade IV cartilage loss on the medial tibial plateau or femoral condyle that potentially could contact a Trammpolin® medial meniscus prosthesis
3. Has lateral compartment pain and Grade III or Grade IV modified Outerbridge cartilage score in the lateral compartment
4. Has a varus or valgus knee deformity of > 5° requiring a tibial or femoral osteotomy
5. Has a varus alignment that is not passively correctable
6. Has a laxity level of more than Grade II (IKDC), primary or secondary to an injury of the anterior cruciate ligament (ACL) and/or posterior cruciate ligament (PCL) and/or lateral collateral ligament (LCL) and/or medial collateral ligament (MCL)
7. Has significant trochlear dysplasia, patellar instability or symptomatic patellar misalignment
8. Has patellar compartment pain and Grade III or Grade IV modified Outerbridge cartilage score in the patellar compartment.
9. Compared to a normal knee, has obvious radiological evidence of medial femoral squaring, anatomical variance in the medial tibial plateau, or irregularly shaped cartilage surface
10. Had an ACL reconstruction performed < 9 months prior to surgery
11. Has a BMI > 30 at the time of screening
12. Has a knee flexion contracture > 10°
13. Has a knee flexion < 90°
14. Had a previous High Tibial Osteotomy (HTO) < 1 year ago
15. Has insufficiency fractures or avascular necrosis of the medial compartment
16. Has an active infection or tumor (local or systemic)
17. Has any type of knee joint inflammatory disease including Sjogren's syndrome
18. Has neuropathic knee osteoarthropathy, also known as Charcot joint
19. Has any medical condition that does not allow possible arthroscopy of the knee
20. Has neurological deficit (sensory, motor, or reflex)
21. Is currently involved in another investigation of the lower extremity
22. Anticipates having another lower extremity surgery during the clinical investigation period
23. Has received any corticosteroid knee injections ≤ 3 months prior to surgery
24. Has proven osteoporosis
25. Is on immunostimulating or immunosuppressing agents
26. Has ipsilateral or contralateral lower limb joint conditions that may affect ambulation or KOOS (e.g. have a leg length discrepancy > 2.5 cm [1 inch], causing a noticeable limp)
27. Is a female who is lactating, expecting, or is intending to become pregnant during the clinical investigation period
28. Is mentally incapacitated (incapable of appraising or controlling conduct) or have mental disability (e.g., dementia or Alzheimer's)
29. Has a condition or be in a situation that, in the Investigator's opinion, may confound the clinical investigation results, may risk the safety of the patient, or may interfere significantly with the subject's participation in the clinical investigation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2021-10-19 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Performance of the Trammpolin® medial meniscus prosthesis | 24 months
  Performance of the Trammpolin® medial meniscus prosthesis in improving pain as assessed by the Knee Osteoarthritis and injury Outcome Score (KOOS) Pain Sub-scale at 24 months post-operative compared to baseline (pre-operative) The minimum value is 0 and maximum value is 100, a score of 100 is being no pain and the highest attainable score

SECONDARY OUTCOMES:
Knee Osteoarthritis and injury Outcome Score (KOOS) Pain | 6 weeks, 3 months, 6 months, 12 months and 24 months
  • Knee Osteoarthritis and injury Outcome Score (KOOS) Pain Sub-scale at 6 weeks, 3 months, 6 months, 12 and 24 months post-operative compared to baseline (pre-operative). A score of 100 is being no pain.
Knee Osteoarthritis and injury Outcome Score (KOOS) overall | at 6 weeks, 3 months, 6 months, 12 months and 24 months post-operative compared to baseline (pre-operative).
  at 6 weeks, 3 months, 6 months, 12 months and 24 months post-operative compared to baseline (pre-operative). A score of 100 is being no pain .
PAIN Visual Analog Scale (VAS) | at 6 weeks, 3 months, 6 months, 12 months and 24 months post-operative
  at 6 weeks, 3 months, 6 months, 12 months and 24 months post-operative compared to baseline (pre-operative). Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between 0 "no pain" and 10 "worst pain"
Lysholm Knee Scoring Scale | at 6 weeks, 3 months, 6 months, 12 months and 24 months
  scale at 6 weeks, 3 months, 6 months, 12 months and 24 months post-operative compared to baseline (pre-operative).
  The Lysholm Knee Scoring Scale consists of eight items that asses: pain, instability, locking, swelling, limp, stair climbing, squatting, and need for support.
  Measurement level per item: mode of scoring (0-25); measurement level ordinal Measurement level total score: mode of scoring (0-100); measurement level ordinal 100 = no symptoms of impairment. Higher scores indicate a better outcome with fewer symptoms or disability.
Oxford Knee Score | at 6, 12 and 24 months
  at 6 months, 12 months and 24 months post-operative compared to baseline (pre-operative).
  The Oxford Knee Score questionnaire consists of 12 questions that cover function and pain of the knee. Each question is scored from 0 to 4 (0 being the worst outcome and 4 being the best). The overall score is the sum of all items and can range from 0 to 48, with higher scores corresponding to better outcomes.
Europol 5D health utility score | at 6, 12 and 24 months
  at 6 months, 12 months and 24 months post-operative compared to baseline (pre-operative).
  Evaluates the generic quality of life, developed in Europe and widely used. Used for estimating QALY to make decisions in resource allocation. The EQ-5D questionnaire has two components: health state description and evaluation. Health state is measured in terms of five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. In the evaluation part, the respondents evaluate their overall health status using the VAS.
Work, Osteoarthritis or joint-Replacement Questionnaire (WORQ) | at 6 weeks, 3 months, 6 months, 12 months and 24 months
  at 6 weeks, 3 months, 6 months, 12 months and 24 months post-operative compared to baseline (pre-operative). The questionnaire consists of 13 items and has a total score from 0 ('very much trouble/ can't do') to 100 ('no trouble at all')
Patient satisfaction on a 5-point Likert scale | at 6 months, 12 months and 24 months
  at 6 months, 12 months and 24 months post-operative compared to baseline (pre-operative).
  The Likert scale consists of a series of statements about a topic, on which the respondent can indicate their level of agreement. For each item, a respondent is asked, using a series of ordered answer options, to indicate the extent to which he agrees with the statement, for example 'totally agree' or 'disagree'. The separate items together indicate the attitude of a respondent towards a subject. The questions uses a 5 or 7 point scale, from one extreme to the other. It is also called a satisfaction scale or satisfaction survey
Knee X-ray (weight-bearing) | 12 months
  To evaluate the height of the joint space compared to baseline (pre-operative).
Knee MRI - Assessment of cartilage condition according to the modified Outerbridge Grading system at screening, 12 and 24 months - Assessment of relative position of the Trammpolin® medial meniscus prosthesis to the tibial plateau | At 12 and 24 months
  Reference 24 CIP: (Jones) Assessment of relative position of the Trammpolin® medial meniscus prosthesis to the tibial plateau, i.e. "extrusion" will be performed according to the method as described by Jones:
  L. D. Jones, S. J. Mellon, N. Kruger, A. P. Monk, A. J. Price, and D. J. Beard, "Medial meniscal extrusion: a validation study comparing different methods of assessment," Knee Surg Sports Traumatol Arthrosc, Apr. 2017, doi: 10.1007/s00167-017-4544-4.
Biopsy of synovium and synovial fluid sample. In case the investigational device requires revision another biopsy is taken from the synovium and a second sample of the synovial fluid. | At implantation and if applicable at explantation
  The baseline samples are stored in the freezer, to be used as baseline values in case the investigational device requires revision during the course of the study. During any secondary surgical procedure, another biopsy is taken from the synovium and a second sample of the synovial fluid. Samples will be compared in a qualitative/descriptive manner according to the method as described by Krenn in PATHOLOGY RESEARCH AND PRACTICE, 2002;198(5):317-25: hyperplasia/enlargement of synovial lining cell layer, inflammatory infiltration, activation of synovial stroma/pannus formation will be assessed. Synovial fluid samples at baseline will be compared to any later sample with respect to the presence and nature of foreign body particles.
Safety of the Trammpolin® medial meniscus prosthesis | 6 weeks, 3 months, 6 months, 12 months and 24 months
  Incidence of adverse events (e.g. hospitalization)
Safety - Incidence of secondary surgery of the index knee | 6 weeks, 3 months, 6 months, 12 months and 24 months
  Incidence of secondary surgery of the index knee

CONTACTS AND LOCATIONS:
Overall Officials: T. van Tienen, MD. PhD., Study Director — Sponsor GmbH
Locations (3):
- Netherlands (3):
  - MUMC+, Maastricht
  - Sint Maartenskliniek, Nijmegen
  - Haaglanden Medisch Centrum, The Hague

IPD SHARING:
Plan to Share IPD: No